CLINICAL TRIAL: NCT02926729
Title: Real-Time Assessment Of Breast Cancer Lumpectomy Specimen Margins With Nonlinear Microscopy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Massachusetts Institute of Technology (Other); Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, James L Connolly, James Connolly, Professor of Pathology, Harvard Medical School; Senior Pathologist Beth Israel Deaconness Medical Center, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16-145
Record Dates: First submitted 2016-10-05; First posted 2016-10-06 (Estimated); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Experimental (Experimental): Standard lumpectomy followed by nonlinear microscopy imaging of excised surgical margins. If invasive cancer or DCIS at or close to the margin is detected, additional excision may be performed.
  Interventions: Device: nonlinear microscopy imaging of excised surgical margins
- Control (Active Comparator): Standard lumpectomy without nonlinear microscopy imaging.
  Interventions: Procedure: standard lumpectomy without nonlinear microscopy imaging

INTERVENTIONS:
Device: nonlinear microscopy imaging of excised surgical margins — Following standard lumpectomy excision, excised tissue will be imaged with NLM. If invasive cancer or ductal carcinoma in situ (DCIS) is detected on or close to the margin, additional excision may be performed. Following surgery, final margins will be evaluated using paraffin embedded histopathology as per standard procedure. Paraffin embedded histopathology will be used to make a final margin determination.
  Arms: Experimental
Procedure: standard lumpectomy without nonlinear microscopy imaging — Lumpectomy with postoperative paraffin embedded histopathology to make a final margin determination.
  Arms: Control

SUMMARY:
This research is studying a new investigative imaging instrument called a nonlinear microscope (NLM). A nonlinear microscope can produce images similar to an ordinary pathologist's microscope, but without first processing tissue to make slides. This study will determine if a NLM can be used to evaluate tissue during lumpectomy surgery for breast cancer in order to reduce the probability that standard pathologic examination of the specimen after the end of the operation will find close or positive margins, thus possibly requiring the patient to have additional breast surgery.

DETAILED DESCRIPTION:
The purpose of this research study is to improve the treatment of breast cancer and reduce the number of patients who require repeat surgical procedures to completely remove breast malignancy.

In standard procedures, pathologists evaluate tissue samples on a microscope after the surgery is over. The new investigative imaging instrument is an advanced type of microscope that enables evaluation during surgery.

The microscope will not be used directly on the participant or in the operating room, but instead will be used to image tissue immediately after excision but prior to the conclusion of surgery. If pathologic examination using NLM concludes that there is invasive cancer or ductal carcinoma in situ (DCIS) at or close to the margin of the specimen, the surgeon will be notified and may decide to do additional surgical shavings before the patient leaves the operating room, in order to improve the likelihood of achieving clean margins and reduce the probability that the patient will be advised to have another operation to achieve clean margins. For both patients on the experimental arm (NLM) and the control arm (without NLM), standard pathologic evaluation of the specimen will be done some days after the lumpectomy is completed. That pathologic evaluation will decide whether or not to recommend that the patient has additional surgery in order to achieve clean margins. The primary outcome measure is the percentage of patients in each group who are advised to have additional surgery for this reason.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled to undergo lumpectomy for breast cancer at BIDMC.
* Core needle biopsy revealing invasive breast cancer or DCIS.
* Female.
* Minimum age of 21 years.
* Eligible for breast conserving surgery, lumpectomy and radiation.
* Estrogen receptor positive (ER+) on core needle biopsy, or if estrogen receptor negative (ER-), have evaluable estrogen receptor status with positive internal control on core biopsy.
* Progesterone receptor positive (PR+) on core needle biopsy if biopsy indicates invasive cancer, or if progesterone receptor negative (PR-) on biopsy indicating invasive cancer, have evaluable progesterone receptor status with positive internal control on core biopsy.
* HER2 IHC and/or FISH ordered on core biopsy, if biopsy indicates invasive cancer.
* Oncotype DX or other genetic assay performed on core biopsy or not requested.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Contraindicated for radiation therapy.
* Pregnancy. (Pregnant women will be excluded from this study because radiation therapy is contraindicated during pregnancy.)
* Current invasive cancer or DCIS at the site of a previous surgery.
* Any systemic neoadjuvant (or preoperative) therapy between the core biopsy and lumpectomy.
* Involvement in another therapeutic trial for breast cancer at Dana Farber or elsewhere.
* Risk of poor cosmetic outcome after initial lumpectomy and possible additional excision, as assessed by a study surgeon.
* Recommendation for mastectomy based on radiology.
* Patients that have complex DCIS as indicated on radiology, which would require excising a large tissue volume.
* No or equivocal ER, PR or HER2 testing performed prior to surgery if biopsy indicates invasive cancer.
* No or equivocal ER testing performed prior to surgery if biopsy indicates ductal carcinoma in situ.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2019-07-17 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Rate of recommendation for repeat surgery on postoperative histopathology | 2 years
  The percent of patients in each arm who have a recommendation for additional surgery because of near or involved margins as a result of the standard postoperative histopathologic review (by a pathologist blinded to whether the patient was on the experimental or control arm).

CONTACTS AND LOCATIONS:
Overall Officials: James Connolly, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No